CLINICAL TRIAL: NCT01613027
Title: A Multicenter Observational Study of the Response to Rituximab (MabThera®) in Seropositive Patients With Rheumatoid Arthritis With Inadequate Response or Intolerance to Treatment With One or More Tumor Necrosis Factor Inhibitors (TNFi)
Brief Title: An Observational Study of MabThera in Participants With Severe Active Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML27998
Record Dates: First submitted 2012-05-25; First posted 2012-06-06 (Estimated); Results first posted 2016-10-24 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Rituximab: Rituximab administered according to prescribing information and normal clinical practice.
  Interventions: Biological: Rituximab

INTERVENTIONS:
Biological: Rituximab — Rituximab administered according to prescribing information and normal clinical practice.
  Other Names: MabThera®

SUMMARY:
This observational study will evaluate the effect on disease activity and the safety in routine clinical practice of MabThera (rituximab) in participants with active seropositive rheumatoid arthritis, who have an inadequate response to one or more tumour necrosis factor inhibitor (anti-TNF) therapies.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years with rheumatoid arthritis (RA)
* Seropositive participants with RA (positive for rheumatoid factor (RF) and/or anti-Citrullinated Cyclic Peptide [CCP])
* Active disease despite receiving one or more TNF inhibitors
* Absence of serious or active infection

Exclusion Criteria:

* Participants with serious history of heart failure (class New York Heart Association [NYHA] IV) or severe uncontrolled heart disease
* Participants pregnant or lactating
* Prior treatment with Mabthera®
* Participants receiving any other investigational product in the context of other clinical study
* Participants with known hypersensitivity to rituximab or to any of the excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with severe active, seropositive rheumatoid arthritis who have an inadequate response or intolerance to anti-TNF therapy
Sampling Method: Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2012-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (8):
- Greece (8):
  - Athens
  - Haidari
  - Heraklion
  - Ioannina
  - Larissa
  - Pátrai
  - Thessaloniki
  - Voula

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rituximab
Started | 135
Completed | 127
Not Completed | 8
Not completed — Lost to Follow-up | 5
Not completed — Switched Physician | 1
Not completed — Lack of Efficacy | 1
Not completed — Patient's Decision Due to Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Intention-to Treat population, defined as all enrolled participants who received at least one dose of rituximab.
Arm/Group | Rituximab
Number analyzed (Participants) | 135
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115
  Male | 20

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Disease Activity Score Based on 28-joint Count and Erythrocyte Sedimentation Rate (DAS28-ESR) at Month 6 and Month 12
Description: DAS28-ESR is a measure of the participant's disease activity and was calculated using the swollen joint count of 28 joints (SJC28), tender joint count of 28 joints (TJC28), erythrocyte sedimentation rate (ESR) (millimeters per hour [mm/hour]) and patient's global assessment of disease activity (100-millimeter [mm] horizontal visual analog scale with 0=no disease activity to 100=maximum disease activity). DAS28-ESR scores range from 0 to 10, with higher scores corresponding to greater disease activity.
Time Frame: Baseline, Month 6, Month 12
Population: Intention-to Treat population, defined as all enrolled participants who received at least one dose of rituximab.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rituximab
Number analyzed (Participants) | 135
units on a scale
  Baseline | 5.53 (1.12)
  Change at Month 6 | -1.52 (1.36)
  Change at Month 12 | -1.88 (1.40)
Statistical Analysis 1: Comparison: Rituximab; Difference in change at Month 6; Test type: Superiority or Other; p < 0.001, Paired t-test
Statistical Analysis 2: Comparison: Rituximab; Difference in change at Month 12; Test type: Superiority or Other; p < 0.001, Paired t-test

2. Secondary Outcome: Percentage of Participants With European League Against Rheumatism (EULAR) Response at Month 6 and Month 12
Description: EULAR response was calculated as the difference between DAS28-ESR scores at baseline and Month 6, and baseline and Month 12, and reported as the percentage of participants with response overall, good response, moderate response, and no response measured at each time point. Good responders = decrease from baseline >1.2 with a DAS28 score of ≤3.2; moderate responders = decrease from baseline >1.2 with a DAS28 score of >3.2, or decrease from baseline >0.6 to ≤1.2 with a DAS28 score of ≤5.1; non-responders = decrease from baseline ≤0.6 or decrease from baseline >0.6 and ≤1.2 with a DAS28 score of >5.1.
Time Frame: Baseline, Month 6, Month 12
Population: Intention-to Treat population, defined as all enrolled participants who received at least one dose of rituximab.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab
Number analyzed (Participants) | 135
percentage of participants
  Overall - Month 6 | 75.6 [67.4 to 82.5]
  Good Response - Month 6 | 45.2 [36.6 to 54.0]
  Moderate Response - Month 6 | 30.4 [22.8 to 38.9]
  No Response - Month 6 | 24.4 [17.5 to 32.6]
  Overall - Month 12 | 77.0 [69.0 to 83.8]
  Good Response - Month 12 | 40.0 [31.7 to 48.8]
  Moderate Response - Month 12 | 37.0 [28.9 to 45.8]
  No Response - Month 12 | 23.0 [16.2 to 31.0]

3. Secondary Outcome: Change From Baseline in Swollen Joint Count (SJC) at Month 6 and Month 12
Description: SJC was determined by examining 28 and 66 joints and identifying when swelling was present. Swelling was recorded on the joint assessment form at baseline, no swelling = 0, swelling =1. The sum of swollen joints, each, ranged from 0 to 28 with 0 as best possible health status and 28 as worst health status. A decrease from baseline indicates improvement.
Time Frame: Baseline, Month 6, Month 12
Population: Intention-to Treat population, defined as all enrolled participants who received at least one dose of rituximab.
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | Rituximab
Number analyzed (Participants) | 135
swollen joints
  Baseline | 6.4 (4.6)
  Change at Month 6 | -3.1 (4.3)
  Change at Month 12 | -3.8 (4.5)

4. Secondary Outcome: Change From Baseline in Tender Joint Count (TJC) at Month 6 and Month 12
Description: TJC was determined by examining 28 and 68 joints and identifying the joints that were painful under pressure or to passive motion. Tenderness was recorded on the joint assessment form at baseline, no tenderness = 0, tenderness = 1. A decrease from baseline indicates improvement.
Time Frame: Baseline, Month 6, Month 12
Population: Intention-to Treat population, defined as all enrolled participants who received at least one dose of rituximab.
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | Rituximab
Number analyzed (Participants) | 135
tender joints
  Baseline | 8.2 (5.5)
  Change at Month 6 | -4.4 (5.3)
  Change at Month 12 | -5.1 (5.3)

5. Secondary Outcome: Change From Baseline in Erythrocyte Sedimentation Rate (ESR) at Month 6 and Month 12
Description: ESR is an direct measure of how much inflammation is in the body. The normal range is 0-22 mm/hour for men and 0-29 mm/hour for women. A decrease from baseline indicates improvement.
Time Frame: Baseline, Month 6, Month 12
Population: Intention-to Treat population, defined as all enrolled participants who received at least one dose of rituximab.
Measure: Mean (Standard Deviation); unit: mm/hour
Arm/Group | Rituximab
Number analyzed (Participants) | 135
mm/hour
  Baseline | 43.1 (23.4)
  Change at Month 6 | -14.1 (22.2)
  Change at Month 12 | -16.3 (24.1)

6. Secondary Outcome: Change From Baseline in C-reactive Protein (CRP) at Month 6 and Month 12
Description: C-reactive protein (CRP) is a blood test marker for inflammation in the body. Normal CRP levels are below 5.0 milligrams per liter (mg/L). A decrease from baseline indicates improvement.
Time Frame: Baseline, Month 6, Month 12
Population: Intention-to Treat population, defined as all enrolled participants who received at least one dose of rituximab. Data at Month 6 and Month 12 are included for participants who had assessments for CRP.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Rituximab
Number analyzed (Participants) | 99
mg/L
  Baseline | 21.8 (39.3)
  Change at Month 6 | -10.7 (34.8)
  Change at Month 12 | -14.1 (38.1)

7. Secondary Outcome: Percentage of Participants Who Remained on Treatment or Discontinued Treatment by Month 6 and Month 12
Time Frame: Up to 12 months
Population: Intention-to Treat population, defined as all enrolled participants who received at least one dose of rituximab.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab
Number analyzed (Participants) | 135
percentage of participants
  Remained on treatment - Month 6 | 93.3
  Discontinued treatment - Month 6 | 6.7
  Remained on treatment - Month 12 | 86.7
  Discontinued treatment - Month 12 | 13.3

8. Secondary Outcome: Reasons for Discontinuation of Treatment by Month 6
Description: Reasons for discontinuation from baseline to Month 6 are presented as the number of participants who discontinued treatment by category of reason for discontinuation.
Time Frame: Baseline to Month 6
Population: Intention-to Treat population, defined as all enrolled participants who received at least one dose of rituximab.
Measure: Number; unit: participants
Arm/Group | Rituximab
Number analyzed (Participants) | 135
participants
  Disease remission | 2
  Lost to follow-up | 2
  Adverse reaction (Allergic reaction) | 1
  Switched physician | 1
  Insurance issues | 1
  Lack of response | 1
  Investigation of reasons for body weight loss | 1

9. Secondary Outcome: Reasons for Discontinuation of Treatment by Month 12
Description: Reasons for discontinuation from baseline to Month 12 are presented as the number of participants who discontinued treatment by category of reason for discontinuation.
Time Frame: Baseline to Month 12
Population: Intention-to Treat population, defined as all enrolled participants who received at least one dose of rituximab.
Measure: Number; unit: participants
Arm/Group | Rituximab
Number analyzed (Participants) | 135
participants
  Disease remission | 3
  Lost to follow-up | 5
  Lack of efficacy | 1
  Lack of response | 1
  Non-satisfactory response | 1
  Adverse reaction (Allergic reaction) | 1
  Adverse reactions (Bradycardia and dermatitis) | 1
  Patient's decision due to adverse event | 1
  Switched physician | 1
  Insurance issues | 1
  Investigation of reasons for body weight loss | 1
  Physician's decision | 1

10. Secondary Outcome: Percentage of Participants With Clinically Meaningful Improvement From Baseline in Modified Health Assessment Questionnaire (M-HAQ)
Description: The M-HAQ is a participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week. Each item scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0 = least difficulty and 3 = extreme difficulty. A negative change from baseline indicates improvement.
  Clinically meaningful improvement was defined as minimum clinically significant reduction from baseline of ≥0.22 at the respective time point.
Time Frame: Up to 12 months
Population: Intention-to Treat population, defined as all enrolled participants who received at least one dose of rituximab. Data for change from baseline at Month 6 and Month 12 are included for participants with available data at each time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab
Number analyzed (Participants) | 135
percentage of participants
  Baseline to Month 6 (n = 89) | 65.9 [57.3 to 73.9]
  Baseline to Month 12 (n = 97) | 71.9 [63.5 to 79.2]

11. Secondary Outcome: Percentage of Participants With Adverse Events (AEs) and Adverse Drug Reactions (ADRs)
Description: An AE was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An ADR was defined as any noxious and unintended response to a medicinal product related to any dose. AEs of special interest includes progressive multifocal leukoencephalopathy (PML), any encephalopathy, hepatitis B or hepatitis B reactivation, gastrointestinal perforation, tuberculosis (TB) or TB reactivation, opportunistic infections, and malignancies.
Time Frame: Up to 12 months
Population: Intention-to Treat population, defined as all enrolled participants who received at least one dose of rituximab.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab
Number analyzed (Participants) | 135
percentage of participants
  Any AE | 37.8
  Any non-serious AE | 32.6
  Any non-serious AE not related to rituximab | 24.4
  Any non-serious ADR | 9.6
  Any serious AE | 6.7
  Any serious AE not related to rituximab | 3.0
  Any serious ADR | 3.7
  Any AE of special interest related to rituximab | 2.2

12. Secondary Outcome: Percentage of Participants With Any Non-Serious AE and Any Serious AE by Intensity
Description: Percentage of participants with any non-serious AE and any serious AE by intensity (mild, moderate, severe) was reported.
  An AE was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: Up to 12 months
Population: Intention-to Treat population, defined as all enrolled participants who received at least one dose of rituximab.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab
Number analyzed (Participants) | 135
percentage of participants
  Any non-serious AE (Mild) | 25.9
  Any non-serious AE (Moderate) | 9.6
  Any non-serious AE (Severe) | 0.0
  Any serious AE (Mild) | 1.5
  Any serious AE (Moderate) | 3.0
  Any serious AE (Severe) | 2.2

13. Secondary Outcome: Percentage of Non-Serious AEs
Description: Percentage of non-serious AEs resolved and ongoing at the time of study completion were reported.
  An AE was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: Up to 12 months
Population: Intention-to Treat population, defined as all enrolled participants who received at least one dose of rituximab.
Measure: Number; unit: percentage of non-serious AEs
Units Other Than Participants: Non-Serious AEs
Arm/Group | Rituximab
Number analyzed (Participants) | 135
Number analyzed (Non-Serious AEs) | 66
percentage of non-serious AEs
  Resolved | 84.8
  Ongoing | 15.2

14. Secondary Outcome: Percentage of Non-Serious ADRs
Description: Percentage of non-serious ADRs at the time of study completion was reported.
  An ADR was defined as any noxious and unintended response to a medicinal product related to any dose.
Time Frame: Up to 12 months
Population: Intention-to Treat population, defined as all enrolled participants who received at least one dose of rituximab.
Measure: Number; unit: percentage of non-serious ADRs
Units Other Than Participants: Non-Serious ADRs
Arm/Group | Rituximab
Number analyzed (Participants) | 135
Number analyzed (Non-Serious ADRs) | 16
percentage of non-serious ADRs | 100.0

15. Secondary Outcome: Percentage of Serious AEs
Description: Percentage of serious AEs resolved and ongoing at the time of study completion was reported.
  An AE was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: Up to 12 months
Population: Intention-to Treat population, defined as all enrolled participants who received at least one dose of rituximab.
Measure: Number; unit: percentage of serious AEs
Units Other Than Participants: Serious AEs
Arm/Group | Rituximab
Number analyzed (Participants) | 135
Number analyzed (Serious AEs) | 9
percentage of serious AEs
  Resolved | 88.9
  Ongoing | 11.1

16. Secondary Outcome: Percentage of Serious ADRs
Description: Percentage of serious ADRs resolved and ongoing at the time of study completion was reported.
  An ADR was defined as any noxious and unintended response to a medicinal product related to any dose.
Time Frame: Up to 12 months
Population: Intention-to Treat population, defined as all enrolled participants who received at least one dose of rituximab.
Measure: Number; unit: percentage of serious ADRs
Units Other Than Participants: Serious ADRs
Arm/Group | Rituximab
Number analyzed (Participants) | 135
Number analyzed (Serious ADRs) | 5
percentage of serious ADRs
  Resolved | 80.0
  Ongoing | 20.0

ADVERSE EVENTS:
Time Frame: Up to 12 months
Description: Safety population, defined as all enrolled participants who received at least one dose of rituximab.
Arm/Group | Rituximab
Serious Adverse Events (participants affected / at risk) | 9/135
Other Adverse Events (participants affected / at risk) | 0/135
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab (N=135)
Bronchitis (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Cerebellar tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Angina pectoris (Cardiac disorders) | 1
Haematocrit decreased (Investigations) | 1
Hip arthroplasty (Surgical and medical procedures) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.